CLINICAL TRIAL: NCT01952353
Title: Efficacy of Preoperative Transarterial Chemoembolization for Resectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis: A Prospective Non-Randomized Comparative Study
Brief Title: Preoperative Transarterial Chemoembolization for Resectable HCC With Portal Venous Invasion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-200602
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Resectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Keywords: Hepatocellular Carcinoma; Transarterial Chemoembolization; Hepatic Resection; Portal Vein Tumor Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy; Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperation TACE arm (Experimental): In the preoperative TACE arm (Arm 2), patients underwent TACE followed by surgical resection. Preoperative TACE sessions were repeated once at 4-week intervals unless patients showed either PD or PVTT PD. Then, the patients were prepared for surgical resection, with the exception of those with unresectable disease after TACE For patients who had unresectable disease after TACE, plans for surgical resection were abandoned and the subsequent treatment course was determined by his/her attending oncologist
  Interventions: Procedure: Preoprative TACE; Procedure: Liver resection plus Thrombectomy
- Resection arm (Active Comparator): Liver resection Plus Thrombectomy
  Interventions: Procedure: Liver resection plus Thrombectomy

INTERVENTIONS:
Procedure: Preoprative TACE
  Other Names: Preoperative transarterial chemoembolization
  Arms: Preoperation TACE arm
Procedure: Liver resection plus Thrombectomy — Liver resection plus Thrombectomy
  Other Names: Removal of all tumor tissue by surgery

SUMMARY:
Whether preoperative transarterial chemoembolization can prolong survival for the resectable hepatocellular carcinoma remains controversial, particularly in patients with portal vein tumor thrombi. This study designs to systematically identify and summarize the effect of preoperative TACE for resectable HCC with portal venous invasion.

DETAILED DESCRIPTION:
With various improvements in interventional radiology, since the 2005 practice guidelines issued by the American Association for the Study of Liver Diseases , transcatheter arterial chemoembolization has become one of the available locoregional therapies for HCC. Transcatheter arterial chemoembolization, which generally performed in intermediate-stage HCC patients, involves injection of an embolizing agent into the hepatic artery to deprive the tumor of its major nutrient source via embolization of the nutrient artery, resulting in ischemic necrosis of the tumor. To prevent intrahepatic recurrence due to portal vein invasion of the HCC tumor, therapeutic strategies such as preoperative TACE, and postoperative adjuvant chemotherapy have been tried. According to the latest and the most powerful evidence, however, preoperative TACE is not routinely recommended for patients undergoing hepatectomy to treat resectable HCC , and TACE may delay surgical treatment or decrease the resection volume of the liver, or it also may create a missed opportunity for surgical treatment.

Rather than subject all these patients to such an invasive procedure and put them at risk for missing opportunity for surgical treatment, it may be better to select optimal candidates to receive surgical resection. Recent studies have even shown favorable long-term survival outcomes of HR in well-selected cases of HCC with PVTT. About whether preoperative transarterial chemoembolization is available for the resectable hepatocellular carcinoma with portal vein tumor thrombi, so far, has hardly been reported.

ELIGIBILITY:
Inclusion Criteria:

* a) age between 18 and 75 years,
* b) HCC with no previous treatment,
* c) the presence of major PVTT or less on imaging,
* d) Eastern Co-operative Group performance status 030 ,
* e) resectable disease

Exclusion Criteria:

* a) Child-Pugh class B or C liver cirrhosis, or evidence of hepatic decompensation including ascites, esophageal or gastric variceal bleeding or hepatic encephalopathy, or ICGR-15 >15%,
* b) an American Society of Anesthesiologists (ASA) score ≥ 3,
* c) the presence of distant metastasis or other malignant diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2006-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
overall survival time | 5years

SECONDARY OUTCOMES:
disease free survival | 5 years
Number of Adverse Events | 30 days
  All severe adverse events for the entire course of treatment, including treatment for primary tumor and recurrent tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- SunYat-sen University cancer center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Peng ZW, Guo RP, Zhang YJ, Lin XJ, Chen MS, Lau WY. Hepatic resection versus transcatheter arterial chemoembolization for the treatment of hepatocellular carcinoma with portal vein tumor thrombus. Cancer. 2012 Oct 1;118(19):4725-36. doi: 10.1002/cncr.26561. Epub 2012 Feb 22. PMID 22359112
- See also: web site of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn